CLINICAL TRIAL: NCT01687556
Title: Epigallocatechin-3-Gallate Improves Acne in Humans by Modulating Intracellular Molecular Targets and Inhibiting P. Acnes
Brief Title: EGCG Improves Acne by Modulating Molecular Targets
Acronym: EGCG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-2005-043-0
Record Dates: First submitted 2010-07-23; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Acne Vulgaris
Keywords: EGCG; green tea
MeSH Terms: conditions — Acne Vulgaris | interventions — Tea; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical EGCG 1% (Active Comparator): Seventeen subjects were designated to use 1% EGCG .Since baseline visits, affected areas of randomly allocated half sides were treated with 1% solution twice daily, whereas those of the opposite sides were treated with vehicle only (3% ethanol).
  Interventions: Other: topical EGCG application on acne
- topical EGCG 5% (Experimental): Eighteen subjects were designated to use 5% EGCG, to evaluate a dose-response relationship. Since baseline visits, affected areas of randomly allocated half sides were treated with 5% EGCG solution twice daily, whereas those of the opposite sides were treated with vehicle only (3% ethanol).
  Interventions: Other: topical EGCG application on acne

INTERVENTIONS:
Other: topical EGCG application on acne — two times application of topical EGCG on acne lesion
  Other Names: Green tea extract, EGCG

SUMMARY:
Epigallocatechin-3-gallate (EGCG) may improve acne vulgaris

* major polyphenolic constituent in green tea
* known as potent anti-carcinogenic, anti-inflammatory, anti-proliferative, and antimicrobial activities
* lipid-lowering and antiandrogenic properties was reported
* EGCG can improve acne vulgaris via one of the above mentioned actions.

DETAILED DESCRIPTION:
Acne vulgaris is one of the most prevalent skin disorders of sebaceous follicles, affecting more than 85% of adolescents in United States. Acne can persist throughout the adulthood, and even a mild form of acne might progress to permanent scarring on the face, chest and back, thereby causing significant physical and psychosocial morbidities. Acne is a multifactorial disease of which etiology has not been fully elucidated, although considerable progress has been made in understanding its pathogenesis during last decade. The major pathogenic features of acne include abnormal ductal keratinization, sebum overproduction, Propionibacterium acnes, and inflammation. Common acne medications such as topical retinoids, antibiotics and isotretinoin are associated with irritation and incomplete responses, increased bacterial resistance or untoward side events, respectively. Thus there is a continuing need for a novel, effective agent targeting different aspects of acne pathogenesis, with minimal side effects.

In the recent decade, epigallocatechin-3-gallate (EGCG), the major polyphenolic constituent in green tea, has attracted much interest on account of its potent anti-carcinogenic, anti-inflammatory, anti-proliferative, and antimicrobial activities. Preclinical, observational, and clinical trial data have indicated that EGCG can inhibit tumor initiation, promotion, progression, and angiogenesis. EGCG also suppresses neutrophil chemotaxis, and has been suggested to improve many diseases that have inflammatory components such as diabetes, kidney injuries, arthritis, allergies, dental caries, cardiovascular, gastrointestinal, and neurodegenerative diseases. In skin, EGCG has been investigated mainly in light of antioxidative, immunopotentiating and anticarcinogenic properties against chemicals or ultraviolet irradiation. Moreover, EGCG has lipid-lowering and antiandrogenic properties, and can downregulate peroxisome proliferator-activated receptor-γ expression. Based on these observations, it can be inferred that EGCG might be effective in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 15 years
* clinical diagnosis of mild to moderate acne vulgaris

Exclusion Criteria:

* known pregnancy or lactation
* any medical illness that might influence the results of the study,
* a previous history of oral acne medication or surgical procedures including laser treatment within 6 month and topical medication within 4 weeks of study enrollment.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Assessment of acne severity | 8 week after baseline
  Lesion counts of non-inflammatory lesions (closed comedone, open comedone) and severity measured by Reeds revised scale

SECONDARY OUTCOMES:
2-mm punch biopsy of acne lesion on the EGCG-treated sides | 8 week after baseline
Standardized clinical photographs | 8 week after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Suh, M.D., Ph.D., Study Director — Department of Dermatology, Seoul National University College of Medicine
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine,, Seoul, South Korea

REFERENCES:
- [Background] Dominguez J, Hojyo MT, Celayo JL, Dominguez-Soto L, Teixeira F. Topical isotretinoin vs. topical retinoic acid in the treatment of acne vulgaris. Int J Dermatol. 1998 Jan;37(1):54-5. doi: 10.1046/j.1365-4362.1998.00254.x. PMID 9522243
- [Background] Abe I, Seki T, Umehara K, Miyase T, Noguchi H, Sakakibara J, Ono T. Green tea polyphenols: novel and potent inhibitors of squalene epoxidase. Biochem Biophys Res Commun. 2000 Feb 24;268(3):767-71. doi: 10.1006/bbrc.2000.2217. PMID 10679280
- [Background] Alexis AF, Jones VA, Stiller MJ. Potential therapeutic applications of tea in dermatology. Int J Dermatol. 1999 Oct;38(10):735-43. doi: 10.1046/j.1365-4362.1999.00796.x. No abstract available. PMID 10561043